CLINICAL TRIAL: NCT01143298
Title: LEO 27847 - A Single Dose Bioavailability Study of Oral Solid Dosage Form Versus Oral Solution Including Fed Versus Fasted State in Healthy Male Subjects
Brief Title: LEO 27847 - Single Dose Bioavailability Study of Oral Solution Versus Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LEO 27847-K01
Record Dates: First submitted 2010-06-01; First posted 2010-06-14 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2010-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LEO 27847 oral solution 0.1 mg (Experimental): LEO 27847 oral solution 0.1 mg
  Interventions: Drug: LEO 27847 oral solution
- LEO 27847 tablet 0.10 mg (Experimental): LEO 27847 tablet 0.10 mg
  Interventions: Drug: LEO 27847 oral solution
- LEO 27847 tablet 0.01 mg (Experimental): LEO 27847 tablet 0.01 mg
  Interventions: Drug: LEO 27847 oral solution

INTERVENTIONS:
Drug: LEO 27847 oral solution

SUMMARY:
The purpose of this phase 1 study is to determine the relative bioavailability following single oral dose administration of LEO 27847 solution compared to LEO 27847 tablets in healthy male subjects as well as to determine the effect of food on the single oral dose pharmacokinetics of LEO 27847 tablets in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions.
* Subjects will be Caucasian males between 18 and 45 years of age, with body mass index (BMI) between 18 and 32 kg/m2 inclusive.
* Subjects will have a minimum weight of 50 kg
* Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations (congenital non haemolytic hyperbilirubinaemia is acceptable)

Exclusion Criteria:

* male subjects who are not willing to use appropriate contraception (such as condom) and for female partners; occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository) from the time of the first dose until 3 months after the final dosing occasion.
* Subjects who have received any prescribed systemic or topical medication within 7 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety
* Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety
* Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety
* Subjects who are still participating in a clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity), or a marketed drug within the past 3 months prior to the first dosing occasion.
* Subjects who have donated any blood, plasma or platelets in the month prior to screening or who have made donations on more than two occasions within the 12 months preceding the first dose administration
* Subjects with a significant history of drug allergy as determined by the Investigator
* Subjects who have any clinically significant allergic disease (excluding non-active hay fever) as determined by the Investigator
* Subjects who have a supine blood pressure and supine pulse rate at screening higher than 140/90 mmHg and 100 beats per minute (bpm), respectively, or lower than 90/50 mmHg and 45 bpm, respectively, confirmed by repeat
* Subjects who consume more than 28 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse as determined by the Investigator
* Subjects who smoke, or who have smoked within 3 months prior to first dose administration
* Subjects with, or with a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological, dermatological or other major disorders as determined by the Investigator
* Subjects who have had a clinically significant illness within 4 weeks of the start of dose administration as determined by the Investigator
* Subjects who are known to have hepatitis, or who are carriers of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody, or who have a positive result to the test for HIV
* Subjects who, in the opinion of their General Practitioner (GP) or the Investigator, should not participate in the study, including subjects suspected for whatever reason of not being able to comply with the requirements of the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
PK parameters | 7 weeks
  AUC and Cmax in each group

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Brooks, MD, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No